CLINICAL TRIAL: NCT05449990
Title: Family Presence on Multidisciplinary Patient Care Rounds in ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Brigitte S. Cypress, EdD, RN, CCRN, ASSOCIATE PROFESSOR, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro2020001614
Record Dates: First submitted 2022-03-28; First posted 2022-07-08 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: control group: 150 patients and one family member experimental group: 150 patients and one family member; 90 healthcare professionals (no intervention, convenience sampling. cross-sectional data collection)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP: survey and Standard Care (SC) (No Intervention): 150 (75 patients and 75 family members)
- EXPERIMENTAL GROUP: participation in patient-and-family-centered interdisciplinary rounds (PFCC-IR) (Experimental): 150 (75 patients and 75 family members)
  Interventions: Other: Participation in PFCC-IR

INTERVENTIONS:
Other: Participation in PFCC-IR — Patient-and-family-centered-care interdisciplinary rounds (PFCC-IR) with the critical care team are standard practice in the ICU but it doesn't usually include family members. The intervention for this study is PFCC-IR that include one family member of the patient.
  Arms: EXPERIMENTAL GROUP: participation in patient-and-family-centered interdisciplinary rounds (PFCC-IR)

SUMMARY:
Family presence on patient care rounds in adult intensive care units remains the least studied area of family-centered care. Despite support from professional organizations and critical care experts, very few critical care units in the United States have written policies allowing family presence (Davidson, 2013). This multidisciplinary prospective, quasi-experimental design study examined if there is a difference in patient and family satisfaction between rounding in the presence of family compared to patient rounding without family members in the adult intensive care unit and determined the nurses' and health care professionals' attitudes toward family presence during multidisciplinary patient care rounds in the ICU of two hospitals. The sample was 150 patients and family members (75 per hospital) and a convenience sampling of 90 healthcare professionals from the two sites. This investigation will have a potential impact on nursing practice and research. Findings obtained from this study may provide further concrete information on the effect of family presence during multidisciplinary patient care rounds, and patient and family satisfaction that will develop policies and standardized approaches to rounding processes that are innovative in diverse critical care settings as well as other non-critical care settings. Data obtained from this research will be used to create patient and family-centered care plans, add new knowledge and educational programs for healthcare professionals

DETAILED DESCRIPTION:
Purpose/Specific Aims The overall goal of this multidisciplinary, multisite quasi-experimental study was to determine whether family presence and engagement during patient-and-family-centered interdisciplinary rounds (PFCC-IR) impacts nurses' and health care professionals' attitudes and patient and family satisfaction with their intensive care unit (ICU) stay. A. Objectives

(1) To examine if there is a difference in patient and family satisfaction between rounding in the presence of family compared to patient rounding without family members in the adult intensive care unit (ICU) using the Patient Satisfaction with Nursing Care Quality Questionnaire ([PSNCQQ], and the Critical Care Family Satisfaction Survey ([CCFSS]; and, (2) To determine ICU nurses' and health care professionals' attitudes toward family presence during PFCC-IR using the Families' Importance in Nursing Care-Nurse's Attitudes ([FINC-NA] scale

B. Hypotheses / Research Question(s) The present study hypothesized that:

H1: There will be greater patient satisfaction when rounding with family present compared to without family present. H2: There will be differences in attitudes towards family presence during PFCC-IR.

Research Design and Methods: This multisite quasi-experimental study was conducted in an adult ICU of two hospitals in southern New Jersey. Approval from the Institutional Review Board (IRB) was obtained before the initiation of the study. Informed consent was obtained from the patients, family members, nurses, and health care professionals. The sample consists of 150 patients and family members (75 dyads per hospital) and 90 healthcare professionals (n = 390 total) that included the ICU Attendings/Intensivists, Fellows, medical residents, respiratory therapists, physical therapists, pharmacists, dietitians and a social worker. Three instruments were used: the FINC-NA, the PSNCQQ, and the CCFSS. The PFCC-IR were led by the ICU Attending or Intensivist. Duration for Study and Each Subject: The patient and family members' participation in the study took 30 minutes to one hour for the rounds, and another 20-30 minutes to complete the survey for an overall total participation time of 2.5 hours.

Sample Size Justification: A sample of 75 dyads or 150 patients and family members was the projected target sample size for this study. Power analysis for the study was calculated based on 80% power to detect a difference, with a significance level of 0.05 (2-tailed), in means of 0.4 with a standard error of 0.8.

Data Collection: All data were collected by the PI after having all subjects signed the informed consent. Family members or significant others attended one to two PFCC-IR on the first week of admission while the patient is in the ICU. The patient questionnaire was given to the patient by the PI to be completed at the time of discharge or within 24 hours of discharge from the ICU.

The family member and/or significant other questionnaires were administered on the day of the patient's discharge from the ICU or within 48 hours of discharge from the ICU. All eligible ICU nurses and health care professionals were given a survey packet by the PI at the beginning and end of the study. Completed questionnaires was returned in a drop box in the ICU.

Consent Procedures: The consent process took place in a private room in the ICU of the hospital. The PI followed-up and scheduled a bedside contact to explain the study fully to the patient during visiting hours or over the telephone.

All questions from subjects were answered by the PI. The patient and family members were given enough time that they need to read and understand the content of informed consent. Informed consents were obtained from all the 390 subjects in this study.

Economic Burden and/or Compensation for Subjects: Subjects did not incur any expenses by participating in this study. No remuneration was given to the subjects.

Risks and Benefits to Subjects: Patients and family members who gave consent participated in the PFCC-IR. No untoward events occurred when the intervention was administered for the whole duration of the study. There are no withdrawal or attrition of subjects.

Current guidelines recommend for families of ICU patients to participate PFCCIR to facilitate patient-family-centered-care. However, there has been relatively little research to inform best practices. Findings obtained from this study may provide further new knowledge on the effect of family presence during PFCCIR, and patient and family satisfaction that will help establish policies and a standardized approach to rounding processes that can be applied, further developed and implemented in different critical care settings as well as other non-critical care settings. Further, it may decrease the ambivalence expressed by diverse health care providers and limit practice variation.

Data Analysis: Data analysis for this study is in progress using the latest version of the SPSS software.

Data Security: Subjects were made aware that they have the right to privacy and that their identities will not be revealed, and the confidentiality of information will be ensured. Identity protection and confidentiality were fully expressed in the consent form. All the data that were collected are stored in a password protected computer located in the researcher's office. Hard copies of transcripts and narratives are stored in a locked cabinet in the researcher's office in the university, to assure safety and preserve the privacy and confidentiality of all participants.

.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the adult ICU over the age of 20 who are awake and alert with a score of above 25 on the Mini-Mental Status (MMS) examination, able to provide informed consent, fill out the questionnaires and who has a family member or significant other who will be willing to participate in the study.
* Family members who are in the patient's primary support system and or caregiver, significant other, or those whom the patient considered or identified as the family who are over the age of 20, able to provide informed consent and will be willing to attend the multidisciplinary rounds while their patient is in the ICU and fill-out the questionnaires.
* All ICU nurses and other health care professionals such as the physicians, respiratory therapists, social workers, and dietitians over the age of 25, male and female nurses, working full time in the ICUs, and willing to provide informed consent will be surveyed.

Exclusion Criteria:

* Any patient with an MMS score below 25 will not be included in the study.
* Patients who are admitted in cardiogenic shock or who are hemodynamically unstable, who are 'intubated' and on mechanical ventilation will be excluded from the study, and with an MMS score of below 20 will be excluded in the study.
* Family members and nurses who are unwilling or will refuse to participate in multidisciplinary rounds will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Assessing Patient Satisfaction Change after Inclusion in patient-and-family-centered rounds using the Patient Satisfaction with Nursing Care Quality Questionnaire (PSNCQQ) scale | Baseline (day 1 when in the study) and post-intervention (4 days after the patient leave the ICU)
  Patient satisfaction with ICU stay was assessed using the Patient Satisfaction with Nursing Care Quality Questionnaire (PSNCQQ) scale. The instrument is a 19-item questionnaire. Cronbach's reliability estimates of 0.97. Participants' responses are provided using a 5-point Likert-type scale. Total possible scores range from 19-95. Lower total scores indicate greater satisfaction with nursing care. The scoring of the scale was: 1 = excellent, 2 = very good, 3 = good, 4 = fair, 5 = poor
Assessing Family Satisfaction Change after Inclusion in patient-and-family-centered rounds using the Critical Care Family Satisfaction Survey (CCFSS) scale | Baseline (day 1 when in the study) and post-intervention(4 days after the patient leave the ICU)
  The 5 subscales of the CCFSS are assurance, proximity, support, comfort, and information. The Cronbach alpha for the total scale was 0.96 and 0.74 - 0.92 for the subscales (Roberti & Fitzpatrick, 2010). When administering the CCFSS, the respondent endorses one of five choices from 1 (very dissatisfied) to 5 (very satisfied) for each of the 20 items. A mean subscale score is calculated for each subscale (range 1 to 5), and a total satisfaction score (range 5 to 25) is computed by summing the five subscale scores. Higher scores for the subscale and total satisfaction scores indicate a greater satisfaction as perceived by a patient's family member (Wasser & Matchett, 2001; Wasser et al., 2001, 2004)
Assessing attitudes of healthcare professionals using the Families' Importance in Nursing Care-Nurse's Attitudes" (FINC-NA), | one time at any point during the study: through study completion, an average of 1 year
  The instrument consists of 26 items and four subscales: families as a resource in nursing care (10 items; score range 10 to 50), family as a conversational partner (8 items, score range 8 to 40), family as a burden ((four items, score range 4 to 20), and family as its own resource ((4 items, score range 4 to 20). Item scores are summed to create a total score that ranges from 26 to 130. After reverse coding negatively worded items from the Fam-B subscale, higher scores indicated more positive attitudes.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte S Cypress, Principal Investigator — Rutgers University School of Nursing Camden
Locations (1):
- Inspira Health Network, Mullica Hill, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results that are and will be reported in published articles based on this study will be available after deidentification (texts, tables, figures, and appendices)
Supporting Information: SAP
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact: brigitte.cypress@rutgers.edu